CLINICAL TRIAL: NCT03303183
Title: Benchmark Ear Impression Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: KEK-ZH Nr.2014-0326
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Ear Anatomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct Ear Scanner (Active Comparator): Digitale impression via direct ear scanner
  Interventions: Device: Direct Ear Scanner
- Silicone Ear impression (Active Comparator): Impression via silicone
  Interventions: Device: Standard Impression technique

INTERVENTIONS:
Device: Standard Impression technique — Silicone impression technique
  Arms: Silicone Ear impression
Device: Direct Ear Scanner — Direct Ear Scanner to scan the ear anatomy
  Arms: Direct Ear Scanner

SUMMARY:
The purpose of this study is to determine the scan quality of the direct ear scanner concerning consistency, accuracy and reliability and to compare the data to common silicone ear impressions by benchmarking the outcome of each impression technique on custom product dummies on participants.

DETAILED DESCRIPTION:
Today's standard for ear impression techniques is the impression taking process with silicone impression material. To use the silicone impression for a hearing aid manufacturing process the geometry of the impression is needed. Modern processes scan the silicone ear impression with specific scanners. Afterwards the digitalized ear impression is uploaded in the modeling software for further proceed. A new ear impression technique is now provided with the direct ear scanner technology. The direct ear scanner can create a digital scan of the outer ear and ear canal. The scan than can directly transferred to the modeling software. The research question of this study is to determine the scan quality of the direct ear scanner concerning consistency, accuracy and reliability and to compare the data to common silicone ear impressions.

ELIGIBILITY:
Inclusion Criteria:

* Only adult participants ≥ 18 years
* Informed consent form as documented by signature
* Ability to fill in a questionnaire conscientious
* Healthy outer ear (Pinna and ear canal, w/o previous surgical procedures)

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Deviation of Direct ear scanner compared to silicone impressions | 1 year
  Deviation of the scan of Direct ear scanner compared to silicone impressions with two viscosities [mm]

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Switzerland